CLINICAL TRIAL: NCT05321173
Title: Non-interventional Feasibility Assessment for Fast-Track Cardiac Anesthesia
Brief Title: Fast-Track in Cardiac Anesthesia
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Eda Balcı, Medical Doctor, Ankara City Hospital Bilkent
Other Study IDs: MH2.6
Record Dates: First submitted 2022-03-23; First posted 2022-04-11 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Cardiac Surgery
Keywords: cardiac anesthesia; fast-track; pandemic; ICU; early recovery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Extubation ≤ 8 hour: Patients who mechanically ventilated less than 8 hours postoperatively
- Extubation > 8 hour: Patients who mechanically ventilated more than 8 hours postoperatively

SUMMARY:
The introduction of fast-track extubation procedures following cardiac surgery has significantly shortened hospitalization times in intensive care units. In this study, it was aimed to determine the obstacles to the early recovery of patients who underwent cardiac surgery in the crisis environment that developed with the pandemic.

DETAILED DESCRIPTION:
After the time we struggled to overcome the many crises that the pandemic period brought to our lives, it has been clearly seen that the decrease in the number of nurses and doctors and the limitation of the number of beds allocated for postoperative intensive care have been mandatory attempts due to the shift of personnel to areas to fight the pandemic. The fact that cardiac surgery operations are not elective and cardiac patients cannot wait for a long time due to their existing pathologies has led physicians to strive to provide the best service with available resources. To ensure that the cardiac surgery operating room and intensive care beds of our hospital can be used more efficiently and to take initiatives to optimize the recovery in the postoperative period are among the important goals of today and the future. The reason for this is not only to reduce costs and loss of workforce but also to be ready for any crisis time. In addition, it is aimed to perform the operations of critical patients without delay and to successfully discharge them. In the postoperative period, if the functions of many basic organ systems can provide the necessary ideal conditions, the patients can be extubated within 8 hours in fast-track cardiac anesthesia (FTCA) programs. Some problems persist or occur in patients with functional problems such as hemodynamics, cardiac, and respiration who do not meet the extubation criteria. For all these reasons, a prospective, cross-sectional study was planned to focus on daily standard practices and improve areas of failure.

Accordingly, this study aimed to examine the preoperative, intraoperative, and postoperative characteristics of patients who underwent cardiac surgery, and to investigate the factors in patients who could not be extubated within 8 hours after surgery.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients who underwent elective or emergency cardiac surgery

Exclusion Criteria:

* Patients undergoing pediatric cardiac surgeries

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who underwent elective or emergency cardiac surgery within 2 months
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
Extubation time | Postoperative period, up to 24 hours
  Mechanical ventilation duration postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: ZELİHA A DEMİR, Professor, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara City Hospital, Ankara, Select State/Province, Turkey (Türkiye)

REFERENCES:
- [Result] Haanschoten MC, van Straten AH, ter Woorst JF, Stepaniak PS, van der Meer AD, van Zundert AA, Soliman Hamad MA. Fast-track practice in cardiac surgery: results and predictors of outcome. Interact Cardiovasc Thorac Surg. 2012 Dec;15(6):989-94. doi: 10.1093/icvts/ivs393. Epub 2012 Sep 5. PMID 22951954
- [Result] Wong WT, Lai VK, Chee YE, Lee A. Fast-track cardiac care for adult cardiac surgical patients. Cochrane Database Syst Rev. 2016 Sep 12;9(9):CD003587. doi: 10.1002/14651858.CD003587.pub3. PMID 27616189
- [Result] Myles PS, Daly DJ, Djaiani G, Lee A, Cheng DC. A systematic review of the safety and effectiveness of fast-track cardiac anesthesia. Anesthesiology. 2003 Oct;99(4):982-7. doi: 10.1097/00000542-200310000-00035. No abstract available. PMID 14508335